CLINICAL TRIAL: NCT05752396
Title: Disrupted Spatial and Temporal Nociceptive Filtering in Adolescents With and Risk for Overlapping Pain Conditions
Brief Title: Overlapping Pain Trajectory Study
Acronym: COPC
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Christopher D. King, Associate Professor, Children's Hospital Medical Center, Cincinnati
Other Study IDs: 2022-0260
Record Dates: First submitted 2023-02-10; First posted 2023-03-02 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Migraine; Musculoskeletal Pain; Functional Abdominal Pain Disorders; Chronic Pain; Widespread Chronic Pain; Low Back Pain; Healthy Volunteers
MeSH Terms: conditions — Migraine Disorders; Musculoskeletal Pain; Chronic Pain; Low Back Pain | interventions — Postsynaptic Potential Summation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic Pain - Localized: Patients with localized pain conditions (n=140)
  Interventions: Other: Conditioned Pain Modulation; Other: Offset Analgesia; Other: Spatial Summation; Other: Temporal Summation
- Chronic Pain - Overlapping: Patients with two or more pain conditions (n=140)
  Interventions: Other: Conditioned Pain Modulation; Other: Offset Analgesia; Other: Spatial Summation; Other: Temporal Summation
- Healthy Participants: Health Participants without a chronic pain condition (n=140)
  Interventions: Other: Conditioned Pain Modulation; Other: Offset Analgesia; Other: Spatial Summation; Other: Temporal Summation

INTERVENTIONS:
Other: Conditioned Pain Modulation — Conditioned pain modulation (CPM) procedure evaluates the change in mechanical and heat pain sensitivity by a contralateral conditioning stimulus (cold immersion). This psychophysical paradigm investigates inhibitory pain modulation processes.
Other: Offset Analgesia — Offset analgesia (OFA) procedure evaluates the disproportionate change in heat pain sensitivity after a slight decrease in stimulus intensity. This psychophysical paradigm investigates inhibitory pain modulation processes.
Other: Spatial Summation — Spatial summation (SS) procedure evaluates the change in heat pain sensitivity when applying two painful stimuli simultaneously compared to one stimulus alone. This psychophysical paradigm investigates facilitatory pain modulation processes.
Other: Temporal Summation — Temporal summation (TS) procedure evaluates the change in mechanical pain sensitivity after exposure to a series of noxious stimuli of the same intensity. This psychophysical paradigm investigates facilitatory pain modulation processes.

SUMMARY:
The goal of this observational study is to learn about spatial and temporal nociceptive filtering in adolescents with chronic overlapping pain conditions (COPCs). The main questions it aims to answer are:

1. If spatial and temporal filtering of nociceptive information is disrupted in youth with COPCs compared with youth with localized pain conditions and healthy controls.
2. If disrupted nociceptive processing at baseline is associated with the transition from a single localized pain condition to COPCs in youth.

Participation includes:

* quantitative sensory testing
* blood draw
* sleep assessment
* questionnaires

DETAILED DESCRIPTION:
While localized primary pain conditions are prevalent in youth, a significant subset of these patients experience multiple pain conditions and meet the criteria for chronic overlapping pain conditions (COPCs). COPCs have a marked negative impact on daily functioning and quality of life in youth and carry a high risk for continued pain and disability into adulthood. The underlying factors contributing to the development and persistence of COPCs in youth are unknown. The current proposal offers an innovative and previously unexplored approach to determine whether disruptions in spatial (concurrent noxious stimuli across the body) and temporal (noxious stimuli presented over time) filtering of nociceptive processing, reflecting pain amplification (e.g., increased facilitation and/or reduced inhibition), contribute to COPCs. Several quantitative sensory testing methods are uniquely positioned to probe disruptions in nociceptive filtering across spatial (spatial summation, SS; conditioned pain modulation, CPM) and temporal (temporal summation, TS; offset analgesia, OFA) domains. Our recent pilot studies found evidence for greater disruptions in spatial (CPM) and temporal (TS) filtering in youth with COPCs. Our primary objective is to determine if spatial and temporal filtering of nociceptive information differentiates youth with COPCs from those with localized pain and healthy controls and determine whether distinct profiles of disrupted nociceptive processing are associated with the transition of localized pain to COPCs. To accomplish this, the current study will leverage expertise and a vast clinical infrastructure (Migraine, Gastroenterology, Rheumatology and Pain Management clinics) at a large pediatric medical center to enroll 140 youth with a localized pain condition (migraine, abdominal pain, local MSK), and 140 youth with COPC's. 140 healthy youth will also recruited to serve as a control group. Following initial phenotyping to delineate disruptions in spatial and temporal dimensions of nociceptive processing (Aim 1), participants will be assessed for changes in pain status (localized to COPCs) every three months for one year (Aim 2). In Aim 1, it is hypothesized that youth with COPCs will show disrupted spatial (reflected by reduced CPM and enhanced SS) and temporal (reflected by enhanced TS and reduced OFA) processing compared to youth with localized pain and healthy controls. These findings will delineate specific disruptions of nociceptive processing in patients with COPCs. For Aim 2, it is hypothesized that a subset of youth with localized pain and disrupted spatial and temporal filtering will develop COPCs. The stability of spatial and temporal filtering will be examined at clinically relevant time points. The investigators will also explore whether other factors, including concomitant treatments, influence the disrupted filtering and the transition to COPCs. Our research will provide the first insight into the presence and impact of disrupted nociceptive filtering related to COPCs and its naturalistic progression from localized pain. This information will be critical in identifying risk patterns that can be useful in the prevention of progression to COPCs and mitigating long-term risk.

ELIGIBILITY:
Inclusion Criteria:

1. General Criteria

   * Access to the internet either by laptop, tablet, or phone (for REDCap Surveys)
   * English-speaking
   * Parent or guardian willing to comply with protocol, complete study assessments, and provide written informed consent
2. Control Specific Criteria

   * No history/active chronic pain
3. Patient Specific Criteria

   * Patients will need a diagnosis of a chronic pain derived congruent with ICD-11 criteria related to headache (migraine, daily headache), abdominal (FAPD), localized MSK (single limb/joint, low back or chest pain), or diffuse MSK (widespread MSK pain)
   * If on medications, they need to be on stable doses of prescribed pain and/or psychiatric medications for 4 weeks before the baseline study visit.

Exclusion Criteria:

1. General Criteria

   * Skin conditions (e.g., eczema) or past skin damage on the arms and legs in or near sites of sensory testing
   * Any comorbid rheumatic disease (e.g., arthritis, lupus), neurological (e.g., epilepsy, traumatic brain injury) or medical condition (e.g., cancer, diabetes)
2. Control Specific Criteria

   * Taking medications that can alter pain sensitivity (e.g., NSAIDs, opioids, stimulants, anticonvulsants; psychiatric)
3. Patient Specific Criteria

   * Present psychiatric disease as defined by DSM IV (e.g. psychosis, bipolar disorder, major depression, generalized anxiety disorder), alcohol or drug dependence, or documented developmental delays or impairments (e.g., autism, cerebral palsy, ADHD, or mental retardation) that, in the opinion of the investigator, would interfere with adherence to study requirements or safe participation in the study

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents with localized and overlapping pain conditions
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Conditioned Pain Modulation (CPM) Profile (Pressure) | Baseline, 3 months, and 12 months
  -CPM is defined by the change in pressure thresholds (increase) before and during cold immersion. Pressure thresholds will be measured using an algometer.
Conditioned Pain Modulation (CPM) Profile (Heat) | Baseline, 3 months, and 12 months
  -CPM is defined by the change in heat pain intensity (decrease) before and during cold immersion. Heat stimuli will be delivered by a thermode and pain intensity measured by participant self report on the visual analog scale.
Offset Analgesia (OA) Profile | Baseline, 3 months, and 12 months
  OFA is defined by the change in heat pain intensity (decrease) after a slight reduction in stimulus intensity (1 Deg C). Heat stimuli will be delivered by a thermode and pain intensity measured continuously during stimuli by participant self report on the computerized visual analog scale.
Temporal Summation (TS) Profile | Baseline, 3 months, and 12 months
  TS is defined by the change in mechanical pain intensity (increase) after exposure to a series of pinprick stimuli. Pain intensity will be measured by participant self report on the visual analog scale.
Spatial Summation (SS) Profile | Baseline, 3 months, and 12 months
  SS is defined by the change (increase) in heat pain intensity between two simultaneously applied thermodes compared to one stimulus thermode only. Pain intensity will be measured by participant self report on the visual analog scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
Discussing options with IRB.

REFERENCES:
- [Background] Coghill RC. The distributed nociceptive system: a novel framework for understanding pain. Scand J Pain. 2022 Sep 22;22(4):679-680. doi: 10.1515/sjpain-2022-0097. Print 2022 Oct 26. PMID 36129140
- [Background] Quevedo AS, Coghill RC. Attentional modulation of spatial integration of pain: evidence for dynamic spatial tuning. J Neurosci. 2007 Oct 24;27(43):11635-40. doi: 10.1523/JNEUROSCI.3356-07.2007. PMID 17959806
- [Background] Quevedo AS, Coghill RC. Filling-in, spatial summation, and radiation of pain: evidence for a neural population code in the nociceptive system. J Neurophysiol. 2009 Dec;102(6):3544-53. doi: 10.1152/jn.91350.2008. Epub 2009 Sep 16. PMID 19759320
- [Background] Nahman-Averbuch H, Schneider VJ 2nd, Chamberlin LA, Kroon Van Diest AM, Peugh JL, Lee GR, Radhakrishnan R, Hershey AD, Powers SW, Coghill RC, King CD. Identification of neural and psychophysical predictors of headache reduction after cognitive behavioral therapy in adolescents with migraine. Pain. 2021 Feb 1;162(2):372-381. doi: 10.1097/j.pain.0000000000002029. PMID 32773592
- [Background] Szikszay TM, Levenez JLM, von Selle J, Adamczyk WM, Luedtke K. Investigation of Correlations Between Pain Modulation Paradigms. Pain Med. 2021 Sep 8;22(9):2028-2036. doi: 10.1093/pm/pnab067. PMID 33587117
- [Background] Maixner W, Fillingim RB, Williams DA, Smith SB, Slade GD. Overlapping Chronic Pain Conditions: Implications for Diagnosis and Classification. J Pain. 2016 Sep;17(9 Suppl):T93-T107. doi: 10.1016/j.jpain.2016.06.002. PMID 27586833
- [Background] Ohrbach R, Sharma S, Fillingim RB, Greenspan JD, Rosen JD, Slade GD. Clinical Characteristics of Pain Among Five Chronic Overlapping Pain Conditions. J Oral Facial Pain Headache. 2020;34(Suppl):s29-s42. doi: 10.11607/ofph.2573. PMID 32975539